CLINICAL TRIAL: NCT04142099
Title: Skin-to-Skin Contact Start Time in Newborns Sucking and Mother's Breastfeeding Willingness and Parent-Infant Attachment Associated
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Principal Investigator, IRB of NTUH Hsin-Chu Branch, National Taiwan University Hospital Hsin-Chu Branch, National Taiwan University Hospital Hsin-Chu Branch
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 107-061-E
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Mother-Child Relationship
Keywords: early maternal and child skin contact, neonatal sucking
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Infant Breastfeeding Assessment Tool Maternal Attachment Inventor Breastfeeding Mothers Social Support Scale Breastfeeding self-efficancy scale-short form
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin to skin contact 60 min group (Experimental): 1. Newborns are exposed to maternal and child skin within five minutes of birth.
  2. Observe the time of newborn spent in suctioning the maternal nipple in 60 minutes of skin to skin contact.
  3. No intervention or forced neonatal suction.
  Interventions: Behavioral: skin to skin contact 60 min group
- skin to skin contact 20 min group (Active Comparator): 1. Newborns are exposed to maternal and child skin within five minutes of birth.
  2. Observe the time of newborn spent in suctioning the maternal nipple in 20 minutes of skin to skin contact.
  3. No intervention or forced neonatal suction.
  Interventions: Behavioral: skin to skin contact 20min group

INTERVENTIONS:
Behavioral: skin to skin contact 60 min group — Newborns are exposed to maternal and child skin within five minutes of birth for 60 min.
  Arms: skin to skin contact 60 min group
Behavioral: skin to skin contact 20min group — Newborns are exposed to maternal and child skin within five minutes of birth for 20 min.
  Arms: skin to skin contact 20 min group

SUMMARY:
The maternal and child skin contact in the early postpartum period, so that the newborn can show effective sucking ability, will affect the self-confidence of the mother's feeding, and is also one of the factors affecting the mother's exclusive breastfeeding. The purpose of this study was to discuss the relationship between the onset of maternal and child skin contact and the relationship between neonatal milk, mother's willingness to breastfeed and parent-child attachment.

DETAILED DESCRIPTION:
To study the design of the mining experiment, the healthy full-term newborn and mother who gave birth by vaginal production in the delivery room of a teaching hospital in a northern region, and the maternal skin joints in the birth of the newborn, calculate the time to start execution, and According to the Infant Breastfeeding Assessment Tool (IBFAT), the time spent on spontaneous sucking behavior of newborns is estimated. The sample is estimated to take 20% sample loss rate. The number of cases received is 52 pairs. For 104 pairs, the researchers first filled 52 pairs of the control group and then received 52 pairs of the experimental group. The control group maintained routine treatment. The experimental group immediately contacted the mother and baby skin within 5 minutes of the birth of the newborn. The maternal and child skin contact process was carried out without forced or non-intervention, 48-72 hours after delivery.

The questionnaire was used to evaluate the mother's breastfeeding self-efficacy, breastfeeding social support, and maternal and child dependence relationships to estimate the difference. The results of the study will be based on the Generalized Estimating Equation (GEE) method to analyze the starting time of different groups of postpartum maternal and child skin contact, different time points for neonatal sucking ability, breastfeeding self-efficacy, breastfeeding social support, maternal and child Dependency changes.

On May 23, 2018, the researcher entered and left with the unit nursing director's promotion and consent, from June 1 to June 11.

In order to avoid interference with the interrogation of the subjects, the control group was first received and the experimental group was received. The control group of the pre-existing study was routine care, and no problems were found. The results of this experimental group showed that after the newborn was born, after 45 minutes of contact with the mother and baby, the milk-seeking reflex could occur and after 5 minutes. As a result of effective sucking, the mother expressed her happiness because of the sucking behavior of the newborn, and was willing to cooperate with the completion of the study to have the reference and basis before the study.

ELIGIBILITY:
Inclusion Criteria:

* 37 weeks to 40 weeks of gestation
* No high risk pregnancy
* No nipple abnormality
* Willing to breastfeed
* Newborn weight 2500-4000 grams

Exclusion Criteria:

* High risk pregnancy
* 37 weeks ago
* Major bleeding during production
* Neonatal life signs abnormality
* Neonatal oral structure abnormalities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
observational skin to skin contact start time in newborns sucking studies | for 20 minute
  observational skin to skin contact start time in newborns sucking studies

SECONDARY OUTCOMES:
observational skin to skin contact start time in newborns sucking studies | for 60 minute
  observational skin to skin contact start time in newborns sucking studies

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Hsin-Chu Branch, Hsinchu
  - National Taiwan University Hospital Hsinchu Branch, Hsinchu

IPD SHARING:
Plan to Share IPD: No